CLINICAL TRIAL: NCT00526838
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of XL228 Administered Intravenously to Subjects With Advanced Malignancies
Brief Title: Study of XL228 Administered Intravenously to Subjects With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL228-002
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Cancer; Lymphoma
Keywords: Solid Tumor; Multiple Myeloma
MeSH Terms: conditions — Neoplasms; Lymphoma; Multiple Myeloma

ARMS (2):
- 1 (Experimental): once-weekly dosing
  Interventions: Drug: XL228
- 2 (Experimental): twice-weekly dosing
  Interventions: Drug: XL228

INTERVENTIONS:
Drug: XL228 — 1-hour IV infusion

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the multi-targeted protein kinase inhibitor XL228 (active against IGF1R, Src, FGFR, and BCR-Abl) administered as a once- or twice-weekly 1-hour intravenous infusion in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a histologically confirmed solid tumor that is metastatic or unresectable, lymphoma, or multiple myeloma, and for which standard curative or palliative measures do not exist or are no longer effective, and there are no known therapies to prolong survival. Subjects treated at the MTD (once-weekly) must have a diagnosis of metastice colorectal carcinoma, relapsed or refractory multiple myeloma, non-small-cell lung cancer (NSCLC), or small cell lung cancer (SCLC). Certain other eligibility requirements must also be met.
* The subject has disease that is assessable by tumor marker, clinical laboratory, physical, or radiologic means.
* The subject is ≥18 years old.
* The subject has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
* The subject has adequate organ and marrow function.
* The subject is capable of understanding the informed consent document and has signed the informed consent document.
* Sexually active subjects (male and female) must use medically acceptable methods of contraception during the course of the study.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening.

Exclusion Criteria:

* The subject has received anticancer treatment (eg, chemotherapy, radiotherapy, cytokines, investigational agent, or hormones) within 14 days before the first dose of study drug.
* The subject has received radiation to >25% of his or her bone marrow within 30 days of treatment with XL228.
* The subject has not recovered to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grade ≤1 from adverse events (AEs) due to investigational or other agents administered more than 14 days prior to study enrollment.
* The subject has a primary brain tumor. Subjects with brain metastases are considered eligible if the subject has not received radiation therapy for brain metastasis within 2 weeks of enrollment and has been on a stable dose of steroids for 2 or more weeks.
* The subject has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, diabetes, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* The subject has a psychiatric illness or social situation that would limit compliance with study requirements.
* The subject is pregnant or breastfeeding.
* The subject is known to be positive for the human immunodeficiency virus (HIV).
* The subject has a known allergy or hypersensitivity to components of the XL228 formulation.
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of XL228 administered as a once-weekly or twice-weekly 1-hour intravenous (IV) infusion in subjects with advanced malignancies. | Assessed at periodic visits
To determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of XL228 administered as a once- or twice-weekly 1-hour IV infusion in subjects with advanced malignancies. | Assessed at periodic visits

SECONDARY OUTCOMES:
To evaluate plasma pharmacokinetics of XL228 administered as a once- or twice-weekly 1-hour IV infusion in subjects with advanced malignancies. | Assessed at periodic visits
To evaluate preliminary safety and efficacy of XL228 when administered at the once-weekly MTD | Assessed at periodic visits

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Michigan Health System, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina